CLINICAL TRIAL: NCT06739174
Title: Three Way Crossover Study: Assessment of Colostomy Bags with an Active Chamber Filter System and Incidence of Filter-Related Complication by People Living with a Colostomy
Brief Title: Assessment of Colostomy Bags with an Active Chamber Filter System and Incidence of Filter-Related Complication
Acronym: BREEZE-01
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Salts Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 24/EE/0241
Record Dates: First submitted 2024-12-09; First posted 2024-12-18 (Actual); Last update posted 2024-12-18 (Actual); Status verified 2024-12

CONDITIONS: Colostomy - Stoma; Colostomy Complications
Keywords: Colostomy bags; Colostomy; Ballooning; Pancaking; Colostomy bag filter-related complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Confidence Be 1-Piece Closed Bag (Active Comparator): The reference device is CE Marked and already commercially available
  Interventions: Device: Confidence Be 1-Piece Closed Bag
- Confidence Natural 1-Piece Closed Bag (Active Comparator): The reference device is CE Marked and already commercially available
  Interventions: Device: Confidence Natural 1-Piece Closed Bag
- Confidence Be go 1-Piece Closed Bag (Active Comparator): The reference device is CE Marked and already commercially available in Australia
  Interventions: Device: Confidence Be go 1-Piece Closed Bag

INTERVENTIONS:
Device: Confidence Be 1-Piece Closed Bag — Active Chamber Filter - Circle Shape
  Arms: Confidence Be 1-Piece Closed Bag
Device: Confidence Natural 1-Piece Closed Bag — Protective Filter - Circle Shape
  Arms: Confidence Natural 1-Piece Closed Bag
Device: Confidence Be go 1-Piece Closed Bag — Active Chamber Filter - Hexagon Shape
  Arms: Confidence Be go 1-Piece Closed Bag

SUMMARY:
This 3-way crossover study aims to evaluate whether colostomy bags with an active chamber filter system reduce the incidence of filter-related complications, such as ballooning and pancaking, help neutralise odour, and minimise faecal leakage through the filter compared to colostomy bags with a protective filter

DETAILED DESCRIPTION:
The study will recruit participants living with a colostomy who experience complications related to colostomy bag filters. The study follows a repeated-measures design, in which each participant will test three types of colostomy bags (A, B, and C) over a 21-day period, divided into three 7-day test periods. During each test period, participants will use one type of colostomy bag for 7-days or up to 21 closed bags. Participants will be instructed to change the colostomy bag as often as they normally would or whenever they deem it necessary

ELIGIBILITY:
Inclusion Criteria:

* Adult aged over 18 years
* Colostomy for 6 months or longer
* Experiences any filter-related complications, such as ballooning, pancaking, odour, or faecal leakage through the filter, at least once a week (7 days)
* Independent in colostomy care
* Using a flat, closed colostomy bag
* Stoma size (diameter) less than 55 mm
* Using a colostomy bag with a hydrocolloid wafer (baseplate)
* Able to read and complete the study questionnaire in English

Exclusion Criteria:

* Uses colostomy irrigation
* Bleeding or broken peristomal skin
* Receiving or had radiotherapy or chemotherapy in the last 2 months
* Pregnant or breastfeeding
* Taking part in another clinical study
* Currently receiving treatment under the care of a stoma clinical nurse specialist

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of ballooning | 21-days
  Evaluation and comparison of the incidence of ballooning in colostomy bags with active chamber filter system and a protective filter

SECONDARY OUTCOMES:
Time of ballooning incidence | 21-days
  Evaluation and comparison of the timing of ballooning over a 24-hour period in colostomy bags with an active chamber filter system and a protective filter
Wear time until ballooning incidence | 21-days
  Evaluation and comparison of the wear time duration of colostomy bags with an active chamber filter system and a protective filter until a ballooning incident occurs
Incidence of pancaking | 21-days
  Evaluation and comparison of the incidence of pancaking in colostomy bags with an active chamber filter system and a protective filter
Time of pancaking incidence | 21-days
  Evaluation and comparison of the timing of pancaking incidents over a 24-hour period in colostomy bags with an active chamber filter system and a protective filter
Wear time until pancaking incidence | 21-days
  Evaluation and comparison of the wear time duration of colostomy bags with active chamber filter system and a protective filter until pancaking incident to occur
Faecal leakage occurrence through the filter | 21-days
  Evaluation and comparison of faecal leakage occurrence through the filter in colostomy bags with an active chamber filter system and a protective filter
Occurrence of odour through the filter | 21-days
  Evaluation and comparison of odour occurrence through the filter in colostomy bags with an active chamber filter system and a protective filter

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Hamson, Principal Investigator — Salt Healthcare
Locations (1):
- Central Skin Sciences Institute (CSSI) Salts Healthcare, Birmingham, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No